CLINICAL TRIAL: NCT01978600
Title: Prospective, Randomized, Single-Center Study to Evaluate 24-hour Intraocular Pressure Control With Brinzolamide 1%/Brimonidine 0.2% Fixed Dose Combination Therapy
Brief Title: Evaluation of Intraocular Pressure Using Simbrinza™ in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M-13-037
Record Dates: First submitted 2013-10-30; First posted 2013-11-07 (Estimated); Results first posted 2015-04-13 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-03

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Open-Angle Glaucoma; Ocular Hypertension; Simbrinza™; Intraocular Pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide; Brimonidine Tartrate; Timolol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SIMBRINZA™ (Experimental): Brinzolamide 1%/Brimonidine 0.2% ophthalmic suspension, 1 drop 3 times a day (8AM, 3PM, 10PM) in each eye for 4 weeks
  Interventions: Drug: Brinzolamide 1%/Brimonidine 0.2% ophthalmic suspension
- Timolol Maleate 0.5% (Active Comparator): Timolol Maleate 0.5%, 1 drop twice a day (8AM, 8PM) in each eye for 4 weeks
  Interventions: Drug: Timolol Maleate 0.5%

INTERVENTIONS:
Drug: Brinzolamide 1%/Brimonidine 0.2% ophthalmic suspension — Commercially marketed and approved for lowering IOP in patients with open-angle glaucoma and ocular hypertension.
  Other Names: SIMBRINZA™
  Arms: SIMBRINZA™
Drug: Timolol Maleate 0.5% — Commercially marketed and approved for lowering IOP in patients with open-angle glaucoma and ocular hypertension.
  Other Names: TIMOPTIC™; TIMOPTIC-XE™; BETIMOL™; ISTALOL™
  Arms: Timolol Maleate 0.5%

SUMMARY:
The purpose of this study is to evaluate intraocular pressure (IOP) over a 24-hour period using Simbrinza™ topical ophthalmic suspension.

DETAILED DESCRIPTION:
This study consisted of two phases, a Screening/Eligibility Phase and a Treatment Phase. Both phases required the patient to complete an overnight stay.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of either open-angle glaucoma or ocular hypertension in both eyes.
* Willing and able to attend all study-related visits and be housed overnight at clinical site for the study assessments.
* Must sign an Informed Consent form.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential if pregnant, breastfeeding, or not using adequate birth control.
* Severe central visual field loss in either eye.
* Chronic, recurrent or severe inflammatory eye disease.
* Ocular trauma or ocular surgery within the past 6 months.
* Ocular infection or ocular inflammation within the past 3 months.
* Clinically significant or progressive retinal disease.
* Other ocular pathology, including severe dry eye, that may in the opinion of the investigator preclude the administration of study medication.
* Any other conditions including severe illness which would make the patient, in the opinion of the Investigator, unsuitable for the study.
* Any medical condition that would preclude the safe administration of a topical beta-blocker.
* Cannot safely discontinue all glucocorticoids administered by any route.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danyel Carr, MS, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 study center located in the US.
Pre-assignment Details: Of the 89 enrolled, 3 participants were exited as screen failures prior to randomization. This reporting group includes all randomized participants (86).
Groups:
- Simbrinza: 1 drop 3 times a day (8AM, 3PM, 10PM) in each eye for 4 weeks
- Timolol: 1 drop twice a day (8AM, 8PM) in each eye for 4 weeks
Period: Overall Study
Arm/Group | Simbrinza | Timolol
Started | 44 | 42
Completed | 44 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Simbrinza | Timolol | Total
Number analyzed (Participants) | 44 | 42 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (10.73) | 59.7 (11.14) | 60.1 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 27 | 51
  Male | 20 | 15 | 35

OUTCOME MEASURES:

1. Primary Outcome: Mean Nocturnal IOP at Week 4
Description: Nocturnal IOP (fluid pressure inside the eye) is the mean of the nocturnal time points assessed (10 PM to 6 AM). IOP was measured with a calibrated applanation tonometer in millimeters of mercury (mmHg). One eye from each subject was chosen as the study eye and only data for the study eye were used for the efficacy analysis. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage).
Time Frame: Week 4: 10PM, 12AM, 2AM, 4AM, 6AM
Population: This analysis population includes all participants who received study medication and had at least one on-therapy study visit.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Simbrinza | Timolol
Number analyzed (Participants) | 44 | 42
mmHg
  Baseline (Day 0) | 24.2 (4.01) | 23.6 (3.31)
  Week 4 | 18.6 (3.61) | 18.9 (2.93)

2. Secondary Outcome: Mean Diurnal IOP at Week 4
Description: Diurnal IOP (fluid pressure inside the eye) is the mean of the diurnal time points assessed (8 AM to 8 PM). IOP was measured with a calibrated applanation tonometer in millimeters of mercury (mmHg). One eye from each subject was chosen as the study eye and only data for the study eye were used for the efficacy analysis. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage).
Time Frame: Week 4: 8AM, 10AM, 12PM, 2PM, 4PM, 6PM, 8PM
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Simbrinza | Timolol
Number analyzed (Participants) | 44 | 42
mmHg
  Baseline (Day 0) | 23.2 (3.17) | 22.2 (2.97)
  Week 4 | 17.3 (3.01) | 17.7 (2.90)

3. Secondary Outcome: Mean 24-hour IOP at Week 4
Description: 24-hour IOP (fluid pressure inside the eye) is the mean of all the time points assessed (8 AM to 6 AM). IOP was measured with a calibrated applanation tonometer in millimeters of mercury (mmHg). One eye from each subject was chosen as the study eye and only data for the study eye were used for the efficacy analysis. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage).
Time Frame: Week 4: 8AM, 10AM, 12PM, 2PM, 4PM, 6PM, 8PM, 10PM, 12AM, 2AM, 4AM, 6AM
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Simbrinza | Timolol
Number analyzed (Participants) | 44 | 42
mmHg
  Baseline (Day 0) | 23.6 (3.30) | 22.8 (2.84)
  Week 4 | 17.9 (3.06) | 18.2 (2.63)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (28 Oct 2013 - 03 Mar 2014). Adverse events were obtained as solicited comments from the study patients and as observations by the Investigator as outlined in the study protocol.
Description: An AE was defined as any untoward medical occurrence in a subject who is administered a study treatment (i.e., initiation of treatment with test article) regardless of whether or not the event has a causal relationship with the treatment. This analysis group includes all participants who received study medication.
Arm/Group | Simbrinza | Timolol
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/42
Other Adverse Events (participants affected / at risk) | 0/44 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.